CLINICAL TRIAL: NCT04049981
Title: Examining Mechanisms of Action in Superpower Glass Behavioral Intervention for Children With Autism
Brief Title: Investigation of Mechanisms of Action in Superpower Glass
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID-19
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Dennis Paul Wall, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 34059; PHIND Dream Team Award (Other: Stanford University); SPARK Pilot Program (Other: Stanford University)
Record Dates: First submitted 2019-08-06; First posted 2019-08-08 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder; Autism
Keywords: digital; autism; mobile health; ASD; mobile therapy; Google Glass; wearable computing; technology
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: 1:1 Randomization
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Facial Engagement (Experimental): This group will receive a version of Superpower Glass that targets specific areas of social deficits associated with autism.
  Interventions: Device: Superpower Glass
- Emotion Recognition (Experimental): This group will receive a version of Superpower Glass that targets different areas of social deficits associated with autism.
  Interventions: Device: Superpower Glass

INTERVENTIONS:
Device: Superpower Glass — The intervention uses the outward-facing camera on the google glasses to read facial expressions and provides social cues within the child's natural environment during usual social interaction and during games accessed via the smartphone application. Participants who receive the Google Glass intervention will be asked to use it for around 20 minutes 3 times a week with their parents.

SUMMARY:
The following study aims to understand the mechanism of action at work in a novel artificial intelligence (AI) tool that runs on Google Glass through an Android app to deliver social emotion cues to children with autism during social interactions. This study will examine 2 versions of software on the Google Glass based wearable intervention system. Participants will receive 1 of 2 versions of the software and use the device at home for 4 weeks. This novel device will use a camera, microphone, head motion tracker to analyze the behavior of the subject during interactions with other people. The system is designed to give participants non-interruptive social cues in real-time and will record social responses that can later be used to help aid behavioral therapy. It is hypothesized that both mechanisms under investigation will contribute to social gains in children over the 4 week period of use.

ELIGIBILITY:
Inclusion Criteria:

* Parent of a child with a professional diagnosis of autism who is at least 18 years old.
* Child with autism is 4-8 years old
* Parent/Guardian is able to drive to Stanford University for 2 in lab appointments.(Lives within driving distance of Stanford University).

Exclusion Criteria:

* Parent/Guardian unable to speak and read in English.
* Child with autism receives Social Communication Questionnaire score>15

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-05-01 (Actual); Study Completion 2020-07-01 (Actual)

PRIMARY OUTCOMES:
Change in socialization subscale scores of the Vineland Adaptive Behavior Scales,3rd Edition (VABS-III) from baseline to week 4. | Baseline (Week 0), Week 4
  Vineland Adaptive Behavior Scales, 3rd edition (VABS-III) Socialization subscale of the Parent/Caregiver Comprehensive form will be administered online to the parents. Scores from the socialization domain of the VABS-III reflects one's functioning in social situations. The socialization subscale is 32 items, where raw scores are converted to IQ-type standard scores--v-scale scores (M=15, SD=3) where scores range from 1 to 24, and factor in age equivalents, growth scale values, and higher scores indicate better adaptive functioning.
Change in Parent Rated Social Responsiveness Scale 2 (SRS-2) from baseline to week 4 | Baseline (Week 0), Week 4
  The Social Responsiveness Scale-2 is a 65-item measure where parents rate their child selecting responses on a Likert Scale. This measure will be used to measure and identify social impairment associated with Autism Spectrum Disorder (ASD) and to quantify its severitySocial Responsiveness Scale (SRS) raw scores measure social abilities with lower scores indicating better social skills. (Raw Score Range: 0 - 195 and T-Score Range: 37- above 90).

SECONDARY OUTCOMES:
Changes in Parent Self Agency Measure scores from Baseline to Week 4 | Baseline (Week 0), Week 4
  The Parent Self Agency Measure (PSAM) is a 5-item measure of parent's overall confidence in their ability to act in the parental role. Where higher scores indicate higher parent self-agency.
Change in ASD symptoms as measured by Brief Observation of Social Communication Change (BOSCC) from baseline to week 4 | Baseline (Week 0), Week 4
  The Brief Observation of Social Communication Change (BOSCC) is designed to measure change in core symptoms of children with autism. It aims to capture change in social communication, interaction, and eye contact. The BOSCC is a semi-structured observation of interaction with parent and experimenter to assess social communication. The test contains 9 items to capture the quality of a child's social interaction, with total scores ranging from 0 to 45, and an additional 3 items to capture restricted repetitive behaviors, with total score of which ranges from 0 to 15. The BOSCC total score consists in the sum of the total score obtained in the first twelve items (ASD specific symptoms), and ranges from 0 to 60, with the three extra items added separately to integrate information. In the total and subscale scores, higher scores correspond to more severe symptoms.

OTHER OUTCOMES:
Stanford-Binet Intelligence Scales, Abbreviated Battery, Fifth Edition (ABIQ) score at baseline | Baseline (Week 0)
  The ABIQ assessment measures a child's IQ based on an abbreviated (10 minute) task that measures Nonverbal Fluid Reasoning and Verbal Knowledge to create a standard score for IQ. It will be completed for each child during Intake. The Area Scores and Test Composite on the Stanford-Binet test have an average score of 100 and a standard deviation of 16. The converted score of the individual being assessed indicates where he/she is relative to the norm. A score exceeding 145 is classified as "Genius or near genius," and scores below 70 are classified as "Borderline deficiency."

CONTACTS AND LOCATIONS:
Overall Officials: Dennis P Wall, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol
Time Frame: Data will become available after subject enrollment and data collection has completed.

REFERENCES:
- See also: Study Recruitment and Information Website — http://autismglass.stanford.edu/
- See also: Wall Lab Website — https://wall-lab.stanford.edu/